CLINICAL TRIAL: NCT03251859
Title: A Randomized, Open-label, Pharmacodynamic and Pharmacokinetic Trial Assessing the Effect of Lowering Ticagrelor Maintenance Dose Early After Myocardial Infarction on Platelet Inhibition (ELECTRA Pilot Study).
Brief Title: Effectiveness of Lower Maintenance Dose of Ticagrelor Early After Myocardial Infarction (ELECTRA) Pilot Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Prof. Jacek Kubica, MD, PhD, Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMUMK202H
Record Dates: First submitted 2017-08-14; First posted 2017-08-16 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Myocardial Infarction
Keywords: platelet reactivity; ticagrelor; myocardial infarction; pharmacodynamics; antiplatelet therapy
MeSH Terms: conditions — Myocardial Infarction | interventions — Ticagrelor

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard ticagrelor maintenance dose (Active Comparator): Ticagrelor 90 mg twice daily for the first 45 days after myocardial infarction treated with percutaneous coronary intervention.
  Interventions: Drug: Ticagrelor 90 mg
- Reduced ticagrelor maintenance dose (Experimental): Ticagrelor 90 mg twice daily for the first 30 days after myocardial infarction treated with percutaneous coronary intervention, then reduction of the maintenance dose to ticagrelor 60 mg twice daily for the next 15 days.
  Interventions: Drug: Ticagrelor 90 mg; Drug: Ticagrelor 60 mg

INTERVENTIONS:
Drug: Ticagrelor 90 mg — Ticagrelor 90 mg twice daily
  Other Names: Brilique 90 mg
Drug: Ticagrelor 60 mg — Ticagrelor 60 mg daily
  Other Names: Brilique 60 mg
  Arms: Reduced ticagrelor maintenance dose

SUMMARY:
The ELECTRA pilot study is a randomized, open-label, pharmacokinetic and pharmacodynamic trial designed to evaluate the effect of ticagrelor maintenance dose reduction on platelet inhibition in stable patients who recently underwent acute myocardial infarction and were treated with percutaneous coronary intervention.

ELIGIBILITY:
Inclusion Criteria:

* provision of informed consent prior to any study specific procedures
* diagnosis of acute ST-segment elevation myocardial infarction or acute non-ST-segment elevation myocardial infarction according to the Third Universal Definition of Myocardial Infarction
* index event treatment with percutaneous coronary intervention
* male or non-pregnant female, aged 18-80 years old

Exclusion Criteria:

* contraindications for ticagrelor
* further coronary revascularization planned during the first 45 days after myocardial infarction
* indications for chronic treatment with oral anticoagulant or low-molecular-weight heparin
* active bleeding
* history of intracranial hemorrhage
* recent gastrointestinal bleeding (within 30 days)
* history of coagulation disorders
* history of moderate or severe hepatic impairment
* history of major surgery or severe trauma (within 3 months)
* active neoplastic disease
* patient requiring dialysis
* chronic inflammatory disease
* current therapy with strong CYP3A inhibitors or strong CYP3A inducers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-08-11 (Actual); Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

PRIMARY OUTCOMES:
Platelet Reactivity Assessed with the VASP assay | 45 days
  Platelet inhibition evaluated with the VASP assay 45 days after myocardial infarction.

SECONDARY OUTCOMES:
Platelet Reactivity Assessed with Multiple Electrode Aggregometry | 45 days
  Platelet inhibition evaluated with Multiple Electrode Aggregometry 45 days after myocardial infarction.
Number of Patients With High Platelet Reactivity according to the VASP assay | 45 days
  Number of Patients With High Platelet Reactivity according to the VASP assay 45 days after myocardial infarction.
Number of Patients With High Platelet Reactivity according to Multiple Electrode Aggregometry | 45 days
  Percentage of Patients With High Platelet Reactivity according to Multiple Electrode Aggregometry 45 days after myocardial infarction.
Plasma concentration of Ticagrelor | 45 days
  Evaluation of ticagrelor plasma concentration 45 days after myocardial infarction.
Plasma concentration of AR-C124910XX | 45 days
  Evaluation of ticagrelor active metabolite plasma concentration 45 days after myocardial infarction.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Jacek Kubica, MD, PhD, Principal Investigator — Collegium Medicum im. Ludwika Rydygiera w Bydgoszczy, Uniwersytet Mikołaja Kopernika w Toruniu; Eliano Navarese, Md, PhD, Principal Investigator — Collegium Medicum, Nicolaus Copernicus University, Bydgoszcz, Poland
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kubica J, Adamski P, Buszko K, Baranska M, Sikora J, Marszall MP, Sobczak P, Sikora A, Kuliczkowski W, Fabiszak T, Kubica A, Jilma B, Alexopoulos D, Navarese EP. Platelet inhibition with standard vs. lower maintenance dose of ticagrelor early after myocardial infarction (ELECTRA): a randomized, open-label, active-controlled pharmacodynamic and pharmacokinetic study. Eur Heart J Cardiovasc Pharmacother. 2019 Jul 1;5(3):139-148. doi: 10.1093/ehjcvp/pvz004. PMID 30689800
- [Derived] Kubica J, Adamski P, Buszko K, Kubica A, Kuliczkowski W, Fabiszak T, Jilma B, Alexopoulos D, Paciorek P, Navarese EP. Rationale and Design of the Effectiveness of LowEr maintenanCe dose of TicagRelor early After myocardial infarction (ELECTRA) pilot study. Eur Heart J Cardiovasc Pharmacother. 2018 Jul 1;4(3):152-157. doi: 10.1093/ehjcvp/pvx032. PMID 29040445